CLINICAL TRIAL: NCT04761913
Title: Investigating Cytokine Storm Biomarkers in Children Presenting to Acute Paediatric Services (Non-intensive Care) With Paediatric Inflammatory Multisystem Syndrome During the Covid-19 Pandemic. An Observation Study
Brief Title: Paediatric Inflammatory Multisystem Syndrome During COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Anglia Ruskin University (Other)
Responsible Party: Sponsor
Other Study IDs: 19/20/048
Record Dates: First submitted 2020-12-11; First posted 2021-02-21 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2021-10

CONDITIONS: Paediatric Inflammatory Multisystem Syndrome Temporally Associated With SARS-Cov-2
Keywords: cytokine storm; biomarkers; PIMS-TS; children; COVID-19
MeSH Terms: conditions — Cytokine Release Syndrome; pediatric multisystem inflammatory disease, COVID-19 related; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During the COVID-19 pandemic, a small minority of children have been presenting to acute paediatric services with a new syndrome, Paediatric Inflammatory Multisystem Syndrome temporally associated with SARS-Cov-2 (PIMS-TS). Children with PIMS-TS present with symptoms of inflammation caused by the immune system going into overdrive - this is likely to be in response to the virus. More severe cases involve inflammation and damage to the heart.

The focus of this project is to identify children with milder forms of PIMS-TS who are at risk of progression to more severe disease. Being able to predict the disease course of PIMS-TS at an early stage is important as it will allow clinicians to decide which patients should be treated with immunosuppressants, which have been shown to reduce the severity of the illness but have side effects.

Early data suggests that children with PIMS-TS have elevated biomarkers associated with an over-reaction of the body's immune system (also known as a 'cytokine storm') reaction. This study will explore whether children presenting with milder PIMS-TS have elevated 'cytokine storm' blood profiles and whether these profiles differ between children who continue to have a mild disease course compared to those who develop severe disease.

DETAILED DESCRIPTION:
During the COVID-19 pandemic a minority of children have presented to acute services with clinical features of a new syndrome known as Paediatric Inflammatory Multisystem Syndrome temporally associated with SARS-Cov-2 (PIMS-TS). This high inflammatory state, likely triggered by the virus, has overlapping features of Kawasaki's and Toxic Shock Syndrome.

The focus of this study is to identify which children presenting with mild PIMS-TS symptoms will go on to develop severe disease requiring intensive care unit (ICU) admission. This is important as data suggests that early aggressive treatment with immunosuppression can lead to a relatively quick resolution in symptoms. The results of this study could allow clinicians to be selective in treating patients in whom the benefits of treatment outweigh the risks.

Early data suggests a 'cytokine storm' is involved in the PIMS-TS disease process. This proposed observational study will investigate whether children presenting to the non-ICU setting with features of PIMS-TS have raised cytokine storm biomarkers and whether these may be used to predict which children go onto develop severe disease.

The proposed study will include up to 15 hospitals across East of England. NHS clinical care teams will identify patients meeting the inclusion criteria and upload anonymised data into a secure web-based study database. Data will be retrieved for retrospective cases from 1st March 2020 and prospective data entered up until September 2021.

One hundred children presenting to acute (non-ICU) paediatric services with symptoms of PIMS-TS during the study period will be included.

The primary objective of the study is to describe the 'cytokine storm' biomarker profiles of children aged between 3 months to 16 years presenting with PIMS-TS to the non-ICU setting, focussing on those biomarkers which are readily accessible to district general hospitals (Pro-Beta Natriuretic peptide [BNP], ferritin, and CRP).

The secondary aims of the study are to:

1. Compare cytokine storm biomarker profiles of children who have a mild disease course to those who develop severe disease to identify whether there are any differences between these groups
2. Evaluate the association between cytokine storm biomarker profiles and severe events
3. Compare i) demographic characteristics (including pre-existing disease), and ii) other routine clinical investigations of children who have a mild disease course and those who develop severe disease to identify any differences between these 2 groups
4. Evaluate the association between vaccination status and disease severity
5. Compare cytokine storm biomarker profiles of children testing positive and those testing negative for SARS-CoV-2 via PCR on 2x nasopharyngeal swabs to identify any differences between these 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Within the age range of 3 months to ≤16 years
* Presenting clinically to non-ICU paediatric acute services at hospitals in the East of England region with symptoms suggestive of PIMS (e.g. incomplete Kawasaki's disease/Toxic Shock Syndrome) i.e. having: persistent fever (>38.0oC for 5 or more days) AND high CRP (>80) AND with one or more of additional features listed in Appendix 1 of the RCPCH document 'Guidance: paediatric multisystem inflammatory syndrome temporarily associated with COVID-19'
* Having either a positive or negative SARS-Cov-2 PCR test

Exclusion Criteria:

* Aged below 3 months old or above 16 years old
* Confirmation of any microbial cause other than SARS-Cov-2 (including bacterial sepsis, staphylococcal or streptococcal shock syndromes, infections associated with myocarditis such as enterovirus). Determination of such microbial causes is by routine testing i.e. blood culture; pneumococcal, meningococcal, group A strep, staph aureus blood PCR; ASOT; EBV, CMV, adenovirus, enterovirus PCR on blood; urine and stool culture; throat swab culture; stool virology.

Ages: 3 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children (aged 3 months to ≤ 16 years) presenting to acute paediatric services (non-ICU) with symptoms of PIMS during the period of the COVID-19 pandemic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Blood biomarker associated with a cytokine storm - Pro-Beta Natriuretic Peptide (measured in pg/mL). | From date of admission to date of discharge from hospital assessed up to 18 months
  Pro-Beta Natriuretic Peptide (BNP) measured as part of routine clinical care. NHS care teams will upload anonymised routine clinical measurements into a secure study database.
Blood biomarker associated with a cytokine storm - Ferritin (measured in µg/L) | From date of admission to date of discharge from hospital assessed up to 18 months
  Ferritin measured as part of routine clinical care. NHS care teams will upload anonymised routine clinical measurements into a secure study database.
Blood Biomarker associated with a cytokine storm - C-Reactive Protein (measured in mg/L) | From date of admission to date of discharge from hospital assessed up to 18 months
  C-Reactive Protein measured as part of routine clinical care. NHS care teams will upload anonymised routine clinical measurements into a secure study database.

SECONDARY OUTCOMES:
Demographic characteristics including age, sex, ethnicity and pre-existing morbidities | At admission to hospital
  Information collected as part of routine clinical care. NHS clinical care teams will upload anonymous data into a secure study database.
Hospital stay data | From date of admission to date of discharge from hospital assessed up to 18 months
  Information collected as part of routine clinical care. NHS clinical care teams will upload anonymous data into a secure study database.
Cytokine storm biomarker measured in mg/L (CRP) | From date of admission to date of discharge from hospital assessed up to 18 months
  Clinical investigations (blood biomarkers) collected as part of routine clinical care
Cytokine storm biomarkers measured in pg/mL (pro-beta natriuretic peptide, IL-6, IFN-gamma, IL-10, TNF-alpha) | From date of admission to date of discharge from hospital assessed up to 18 months
  Clinical investigations (blood biomarkers) collected as part of routine clinical care
Full blood count measures in 10^9/L (white cell count - neutrophil and lymphocyte count and platelet) | From date of admission to date of discharge from hospital assessed up to 18 months
  Clinical investigations (blood biomarkers) collected as part of routine clinical care
Full blood count measures in L/L (haematocrit) | From date of admission to date of discharge from hospital assessed up to 18 months
  Clinical investigations (blood biomarkers) collected as part of routine clinical care
Haemoglobin in g/L or g/dL (measured as part of full blood count and blood gas analysis) | From date of admission to date of discharge from hospital assessed up to 18 months
  Clinical investigations (blood biomarkers) collected as part of routine clinical care
Blood gas analysis measured in KPa (pCO2, pO2) | From date of admission to date of discharge from hospital assessed up to 18 months
  Clinical investigations (blood biomarkers) collected as part of routine clinical care
Blood gas analysis measured in mmol/l (glucose, lactate, Na, K and Cl) | From date of admission to date of discharge from hospital assessed up to 18 months
  Clinical investigations (blood biomarkers) collected as part of routine clinical care
Blood gas analysis measured in mmol/l or mEq/L (HCO3, BE) | From date of admission to date of discharge from hospital assessed up to 18 months
  Clinical investigations (blood biomarkers) collected as part of routine clinical care
Liver function tests measured in g/L (protein, albumin, globulin) | From date of admission to date of discharge from hospital assessed up to 18 months
  Clinical investigations (blood biomarkers) collected as part of routine clinical care
Liver function tests measured in U/L (ALP/ALT) | From date of admission to date of discharge from hospital assessed up to 18 months
  Clinical investigations (blood biomarkers) collected as part of routine clinical care
Liver function tests measured in µmol/L (bilirubin) | From date of admission to date of discharge from hospital assessed up to 18 months
  Clinical investigations (blood biomarkers) collected as part of routine clinical care
Troponin measured in ng/ml or ng/L | From date of admission to date of discharge from hospital assessed up to 18 months
  Clinical investigations (blood biomarkers) collected as part of routine clinical care
vitamin D measured in nmol/L | From date of admission to date of discharge from hospital assessed up to 18 months
  Clinical investigations (blood biomarkers) collected as part of routine clinical care
Amylase, CK, LDH measured in U/L | From date of admission to date of discharge from hospital assessed up to 18 months
  Clinical investigations (blood biomarkers) collected as part of routine clinical care
Glucose and triglycerides measured in mmol/L | From date of admission to date of discharge from hospital assessed up to 18 months
  Clinical investigations (blood biomarkers) collected as part of routine clinical care
Urea and electrolytes measured in mmol/L (Na, K, urea) | From date of admission to date of discharge from hospital assessed up to 18 months
  Clinical investigations (blood biomarkers) collected as part of routine clinical care
Urea and electrolytes measured in µmol/L (creatinine) | From date of admission to date of discharge from hospital assessed up to 18 months
  Clinical investigations (blood biomarkers) collected as part of routine clinical care
ferritin measured in µg/L | From date of admission to date of discharge from hospital assessed up to 18 months
  Clinical investigations (blood biomarkers) collected as part of routine clinical care
fibrinogen measured in g/L | From date of admission to date of discharge from hospital assessed up to 18 months
  Clinical investigations (blood biomarkers) collected as part of routine clinical care
D-dimer measured in ng/ml | From date of admission to date of discharge from hospital assessed up to 18 months
  Clinical investigations (blood biomarkers) collected as part of routine clinical care
PT and APTT measured in seconds | From date of admission to date of discharge from hospital assessed up to 18 months
  Clinical investigations (blood biomarkers) collected as part of routine clinical care
INR as a ratio (Patient PT/Control PT) | From date of admission to date of discharge from hospital assessed up to 18 months
  Clinical investigations (blood biomarkers) collected as part of routine clinical care
Acute Kidney Injury graded as no AKI or stage of AKI (1-3) | From date of admission to date of discharge from hospital assessed up to 18 months
  Clinical investigations (blood biomarkers) collected as part of routine clinical care
Positive or negative COVID-19 antibody test | From date of admission to date of discharge from hospital assessed up to 18 months
  Clinical investigations (blood biomarkers) collected as part of routine clinical care
Presence or absence of clinical conditions as assessed by ECG/echocardiography | From date of admission to date of discharge from hospital assessed up to 18 months
  Conditions will include: myocarditis, valvulitis, pericardial effusion, coronary artery dilation, or other conditions.
Presence or absence of clinical conditions as assessed by chest x-ray/chest CT | From date of admission to date of discharge from hospital assessed up to 18 months
  Conditions will include: presence of patchy symmetrical infiltrates, pleural effusion, coronary artery abnormalities (CT with contrast) or other conditions.
Presence or absence of clinical conditions as assessed by abdominal ultrasound | From date of admission to date of discharge from hospital assessed up to 18 months
  Conditions will include: colitis, ileitis, lymphadenopathy, ascites, hepatosplenomegaly or other conditions.
Proteinuria as assessed by urinalysis graded as no protein, protein ++ or protein +++ | From date of admission to date of discharge from hospital assessed up to 18 months
Positive or negative COVID swab result as assessed by PCR | From date of admission to date of discharge from hospital assessed up to 18 months
Positive or negative NPA or throat swab result for respiratory panel as assessed by PCR | From date of admission to date of discharge from hospital assessed up to 18 months
  Including: pneumococcal, meningococcal, Group A Strep, Staph Aureus, EBV, CMV, Andenovirus, Enterovirus
Vaccination status | At admission to hospital
  Information collected as part of routine clinical care. NHS clinical care teams will upload anonymous data into a secure study database.

CONTACTS AND LOCATIONS:
Overall Officials: Jo-Anne Johnson, MRCPCH, PhD, Principal Investigator — Anglia Ruskin University
Locations (6):
- United Kingdom (6):
  - Mid Essex Hospital Trust, Chelmsford, Essex
  - East Suffolk and north Essex NHS Foundation Trust, Colchester, Essex
  - The Princess Alexandra Hospital NHS Trust, Harlow, Essex
  - James Paget University Hospitals NHS Foundation Trust, Great Yarmouth, Norfolk
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk
  - East Suffolk and North Essex Foundation Trust, Ipswich, Suffolk